CLINICAL TRIAL: NCT02647632
Title: Study to Assess Efficacy and Safety of Grazoprevir/Elbasvir Associated With Sofosbuvir and Ribavirin in HCV Genotype 1 or 4-infected Patients Who Failed Direct Acting Antivirals (DAA) Bitherapy With Sofosbuvir
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANRS HC34 REVENGE
Record Dates: First submitted 2015-12-16; First posted 2016-01-06 (Estimated); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Hepatitis C
Keywords: HCV genotype 1 or 4; failure to DAA
MeSH Terms: conditions — Hepatitis C | interventions — elbasvir-grazoprevir drug combination; grazoprevir; Sofosbuvir; Ribavirin

ARMS (2):
- 16 weeks of treatment (Experimental): Drug : Grazoprevir/Elbasvir + Sofosbuvir + Ribavirin during 16 weeks
  Interventions: Drug: Grazoprevir/Elbasvir; Drug: Sofosbuvir; Drug: Ribavirin
- 24 weeks of treatment (Experimental): Drug : Grazoprevir/Elbasvir + Sofosbuvir + Ribavirin during 24 weeks
  Interventions: Drug: Grazoprevir/Elbasvir; Drug: Sofosbuvir; Drug: Ribavirin

INTERVENTIONS:
Drug: Grazoprevir/Elbasvir
  Other Names: Grazoprevir/Elbasvir is also known as MK-5172A or Zepatier
Drug: Sofosbuvir
  Other Names: Sofosbuvir is also known as Sovaldi
Drug: Ribavirin
  Other Names: Ribavirin is also known as Rebetol

SUMMARY:
The primary objective of this study is to estimate, in HCV genotype 1 or 4-infected patients who failed a prior DAA bitherapy with Sofosbuvir, the efficacy of a treatment with Grazoprevir/Elbasvir, Sofosbuvir and Ribavirin in the two treatment groups and compare the rate of sustained virological response (SVR) 12 weeks after 16 or 24 weeks of this treatment. SVR12 is defined as HCV RNA < LLOQ (either TD[u] or TND).

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥18 years
* Infection with HCV genotype 1 or 4, confirmed by detectable HCV RNA at pre-inclusion
* Failure to a prior therapy with Sofosbuvir +/- Ribavirin associated with Simeprevir or Daclatasvir or Ledipasvir, with documented presence of NS5A or NS3/4A RAVs (Resistance Associated Variants) at the time of failure (presence of RAVs on at least one sample since the time of failure).

The proportion of patients previously treated with Simeprevir will be limited to a third of all patients included.

* Fibrosis at any stage
* Men and women of child-bearing age and their heterosexual partners must use adequate contraceptions from 15 days before their inclusion in the study up to 7 months after the end of treatment for men and up to 4 months after the end of treatment for women
* Written informed consent signed by the patient and the investigator (on the day of the pre-inclusion at the latest and before any examination required by the study) (article L1122-1-1 Public Health Code)
* Patients with Health insurance (Sécurité Sociale or Couverture Médicale Universelle)

Exclusion Criteria:

* Child B or C cirrhosis (or Child A patients with history of Child B)
* Patients with documented presence of RAVs conferring resistance to sofosbuvir
* Positive HBs Antigen
* Confirmed HIV-1 or HIV-2 infection
* Pregnant or breast-feeding women or men whose female partners are pregnant
* Transplant recipients
* Any evolutive ongoing malignant disease, including hepatocellular carcinoma, which will be specifically screened for before inclusion
* History of severe rhythm disorders or cardiac disease (coronary artery disease, heart failure, arteriopathy,…): the opinion of a cardiologist is compulsory (< 6 months)
* Consumption of alcohol which, in the investigator's opinion, will be an obstacle to the patient's participation and to his/her remaining in the study
* Drug addiction which, in the investigator's opinion, will be an obstacle to the patient's participation and to his/her remaining in the study. Patients included in a programme of substitution with methadone or buprenorphine could be included. The opinion of an addictology consultant is recommended for patients presenting with current drug use or drug use in the past year
* Patients taking part in another clinical trial within 30 days prior to inclusion
* Patient under guardianship, trusteeship or judicial protection

Non-inclusion biological criteria

* Hemoglobin < 11 g/dL
* Platelets < 50 000/mm3
* INR > 1.5 unless subject has known hemophilia or is stable on an anticoagulant regimen affecting INR
* ALT or AST > 10xULN
* Creatinine clearance < 50 mL/mn (MDRD formula)
* Albumin < 30 g/L
* HbA1c > 10% (only in diabetic patients)

Criteria related to study drugs

* Contra-indication to treatment with Grazoprevir/Elbasvir, Sofosbuvir or Ribavirin including a history of hypersensitivity to one of their excipients
* Patients with a non-compliance history, who will be at risk of not complying with the study follow-up timetable
* Treatment with contra-indicated associated drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-01; Primary Completion 2017-01 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
rate of the Sustained Virological Response 12 weeks after the end of the therapy (SVR12), i.e. at W28 or W36 for treatment duration of 16 weeks and 24 weeks respectively. | Week 28 (W28) or Week 36 (W36)
  The primary endpoint is the rate of the Sustained Virological Response defined as HCV RNA < LLOQ (either TD[u] or TND) 12 weeks after the end of the therapy associating Grazoprevir/Elbasvir, Sofosbuvir and Ribavirin (SVR12), i.e. at W28 or W36 for treatment duration of 16 weeks and 24 weeks respectively.

SECONDARY OUTCOMES:
SVR rate 4 weeks after the end of treatment (i.e. at week 20 or week 28 for treatment duration of 16 weeks and 24 weeks respectively) and 24 weeks after the end of treatment (i.e. at week 40 or week 48). | Week 20 (W20) or Week 28 (W28), and W40 or W48
HCV viral load assessment | from Day 0 (D0) to Week 40 (W40) or Week 48 (W48)
Assessment of HCV subtypic distribution at baseline | Pre-inclusion
Numbers and proportions of patients presenting variants of resistance (RAV) at baseline | Pre-inclusion
  The numbers and proportions of patients presenting variants of resistance (RAV) and their characteristics will be studied
Assessment of liver fibrosis by Hepatic impulse elastometry (Fibroscan®), or biological parameters (FibroMeter® or Fibrotest®) | Pre-inclusion, Week 40 or Week 48
For cirrhotic patients, description of the risk of cirrhosis evolution (decompensation, hepatocarcinoma) | Pre-inclusion, Day 0 (D0), Week 16 (W16), W20, W24, W28, W36, W40 or W48
  Cirrhosis evaluation (Child-Pugh)
For cirrhotic patients, description of the risk of cirrhosis evolution (decompensation, hepatocarcinoma) | Pre-inclusion, Day 0 (D0), Week 16 (W16), W20, W24, W28, W36, W40 or W48
  Cirrhosis evaluation (MELD score)
Clinical and biological adverse events occurring during the treatment and until 24 weeks after the end of the treatment | from Day 0(D0) to Week 40 (W40) or W48
Numbers and proportions of patients who interrupted the treatments of the study | from Day 0 (D0) to Week 40 (W40) or W48
Patient's reported outcomes evaluation with questionnaires | Day 0 (D0), Week 4 (W4), W16, W28, W40 or D0, W4, W16, W24, W36, W48 (24 weeks treatment-arm))
  Evaluation of patient's quality of life
Patient's reported outcomes evaluation with questionnaires | Day 0 (D0), Week 4 (W4), W16, W28, W40 or D0, W4, W16, W24, W36, W48 (24 weeks treatment-arm))
  Evaluation of perceived symptoms (ANRS questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Victor DE LEDINGHEN, Principal Investigator — Hôpital de Haut-Lévêque, CHU de Bordeaux; Eric BELLISSANT, Study Chair — Centre de Méthodologie et de Gestion, CHU de Rennes

REFERENCES:
- [Derived] de Ledinghen V, Laforest C, Hezode C, Pol S, Renault A, Alric L, Larrey D, Metivier S, Tran A, Jezequel C, Samuel D, Zoulim F, Tual C, Pailhe A, Gibowski S, Bourliere M, Bellissant E, Pawlotsky JM. Retreatment With Sofosbuvir Plus Grazoprevir/Elbasvir Plus Ribavirin of Patients With Hepatitis C Virus Genotype 1 or 4 Who Previously Failed an NS5A- or NS3-Containing Regimen: The ANRS HC34 REVENGE Study. Clin Infect Dis. 2018 Mar 19;66(7):1013-1018. doi: 10.1093/cid/cix916. PMID 29077864